CLINICAL TRIAL: NCT02538731
Title: Randomized Trial of Spyglass Guided Laser Lithotripsy Versus Dilation-Assisted Stone Extraction for the Endoscopic Removal of Difficult Large Bile Duct Stones
Brief Title: Laser Lithotripsy for Difficult Large Bile Duct Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, guodong li, guodong li, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sdqfs001
Record Dates: First submitted 2015-08-30; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Sphincterotomy, Endoscopic; Cholangiopancreatography, Endoscopic Retrograde; Lithotripsy, Laser

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dilation-assisted group (Other): Dilation-assisted group:Dilation-assisted stone extraction
  Interventions: Procedure: dilation-assisted stone extraction
- laser lithotripsy group (Other): laser lithotripsy group:laser lithotripsy
  Interventions: Device: Spyglass Guided Laser Lithotrips

INTERVENTIONS:
Procedure: dilation-assisted stone extraction
  Arms: Dilation-assisted group
Device: Spyglass Guided Laser Lithotrips
  Arms: laser lithotripsy group

SUMMARY:
Very large bile duct stones are difficult to remove. Dilation-assisted stone extraction, also termed small endoscopic sphincterotomy plus endoscopic papillary large balloon dilatation, is safe and effective technique for the treatment of large CBD stones. However, in approximately 5-10% of patients, the removal of large bile duct stones may be difficult. For this selected group of patients for whom all conventional endoscopic stone treatment devices have failed, laser lithotripsy technology has provided an approach to the fragmentation of difficult bile duct stones.

A single-operator cholangioscopy (SOC) system (SpyGlass Direct Visualization System, Boston Scientific Corp., Natick, MA, USA) has overcome most of the conventional cholangioscopy limitations. The investigators aimed to evaluate the efficacy and safety of Spyglass-guided laser lithotripsy for difficult CBD stones not amenable to conventional dilation-assisted stone extraction therapy.

DETAILED DESCRIPTION:
Purpose Very large bile duct stones are difficult to remove.Dilation-assisted stone extraction, also termed small endoscopic sphincterotomy plus endoscopic papillary large balloon dilatation, is safe and effective technique for the treatment of large CBD stones.However, in approximately 5-10% of patients, the removal of large bile duct stones may be difficult. For this selected group of patients for whom all conventional endoscopic stone treatment devices have failed, laser lithotripsy technology has provided an approach to the fragmentation of difficult bile duct stones.

A single-operator cholangioscopy (SOC) system(SpyGlass Direct Visualization System, Boston Scientific Corp., Natick, MA, USA) has overcome most of the conventional cholangioscopy limitations.We aimed to evaluate the efficacy and safety of Spyglass-guided laser lithotripsy for difficult CBD stones not amenable to conventional dilation-assisted stone extraction therapy.

Study Type: Interventional Study Design: Allocation: Randomized Endpoint Classification: Safety/Efficacy Study Intervention Model: Parallel Assignment Masking: Single Blind (Subject) Primary Purpose: Treatment Official Title: Randomized Trial of Spyglass Guided Laser Lithotripsy Versus Dilation-Assisted Stone Extraction for the Endoscopic Removal of Difficult Large Bile Duct Stones

Primary Outcome Measures:

• Bile Duct Stone Clearance Confirmation that no further stones remain in the bile duct of the patient by cholangiography. Additionally, serum laboratory abnormalities in AST, ALT, Alkaline Phophatase, or bilirubin, or epigastric abdominal pain attributable to bile duct stones.

Secondary Outcome Measures:

* Number of ERCP
* The number of ERCP procedures required to complete clearance of bile duct stones.
* Total Procedure Time
* The total time in minutes for all the ERCP procedures required for stone removal.
* Estimated Procedure Cost
* The cost of patient management for bile duct stones based on the cost of the procedure, hospitalization, and associated costs of complications of cholangitis, pancreatitis, perforation, and bleeding.
* Cholangitis Cholangitis after or between ERCP procedures will be defined as a presentation with epigastric abdominal pain, temperature greater than 38.5 Celsius accompanied by either laboratory abnormalities of the AST, ALT, Alkaline Phosphatase, or Bilirubin or abnormal imaging of the biliary tree on ultrasound,computed tomography scan, or magnetic resonance cholangiopancreatography.
* Pancreatitis
* Pancreatitis following or between ERCP procedures will be defined as the onset of epigastric abdominal pain and either amylase or lipase greater than 3 times the upper limit of normal or findings on ultrasound, computed tomography scan, or magnetic resonance cholangiopancreatography suggestive of pancreatic inflammation.
* Bleeding
* Bleeding attributable to stone therapy will be defined as a drop in hemoglobin by more than 1 gm/dl following or between ERCP procedures with no other cause identified on standard clinical evaluation.

Eligibility

Ages Eligible for Study: 18 Years and older Genders Eligible for Study: Both Accepts Healthy Volunteers: No Criteria

Inclusion Criteria:

• Bile duct stone >1.5cm demonstrated on ultrasound, computed tomography, or magnetic resonance imaging

Exclusion Criteria:

* Biliary, gallbladder or pancreatic malignancy
* Pregnant
* Prior biliary diversion surgery
* Under age 18
* Unable to give informed consent

ELIGIBILITY:
Inclusion Criteria:

* Bile duct stone >1.5cm demonstrated on ultrasound, computed tomography, or magnetic resonance imaging

Exclusion Criteria:

* Biliary, gallbladder or pancreatic malignancy
* Pregnant
* Prior biliary diversion surgery
* Under age 18
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Bile Duct Stone Clearance | 1 hour